CLINICAL TRIAL: NCT00949013
Title: Evaluation of the Expression of the Cancer Stem Cell Marker ALDH1 as a Predictor of Adjuvant Chemotherapy Response in Breast Cancers of High Risk Women in SWOG-9313
Brief Title: S9313B Study of Tumor Tissue Samples From Women With Early-Stage Breast Cancer Enrolled on Clinical Trial SWOG-9313
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000632885; S9313B-ICSC (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Immunohistochemistry

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients enrolled on clinical trial SWOG-9313 will respond to doxorubicin and cyclophosphamide.

PURPOSE: This laboratory study is looking at tumor tissue samples from women with early-stage breast cancer enrolled on clinical trial SWOG-9313.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if ALDH1 positivity, as determined by IHC staining, identifies a poor prognostic subgroup of women with early-stage breast cancer who have been uniformly treated with adjuvant doxorubicin and cyclophosphamide on clinical trial SWOG-9313.

Secondary

* To determine associations of ALDH1 expression with other known factors that have been determined on clinical trial SWOG-9313, such as estrogen receptor (ER) status, HER2 status, TOPOII, cyclin E, and p27.
* To determine if ALDH1 positivity, as determined by IHC staining, identifies a poor prognostic subgroup within ER and HER2 subgroups in patients treated on clinical trial SWOG-9313.

OUTLINE: This is a multicenter study.

Tumor tissue samples from clinical trial SWOG-9313 are analyzed for ALDH1 expression by IHC.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Tumor samples collected from women diagnosed with early-stage breast cancer on clinical trial SWOG-9313 available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled to S9313 consenting to banking
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Correlation of ALDH1 with disease-free survival and overall survival | Retrospectively

SECONDARY OUTCOMES:
Correlation of ALDH1 with other biomarkers (TOPOII, HER2, ER, PgR) | Retrospectively

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F. Hayes, MD, Study Chair — University of Michigan Rogel Cancer Center